CLINICAL TRIAL: NCT00670202
Title: The Effect of Fasudil on Rho Kinase Activity in Patients Scheduled for Elective Carotid Endarterectomy
Brief Title: Rho Kinase (ROCK) Inhibition in Carotid Atherosclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Anju Nohria, Associate Physician in Internal Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P-002369
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Carotid Stenosis
Keywords: Patients scheduled for elective carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis | interventions — fasudil

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, parallel arm design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Fasudil hydrochloride (Experimental): Fasudil hydrochloride 40 mg three times a day X 14 days
  Interventions: Drug: Fasudil Hydrochloride
- Drug: Placebo oral tablet (Placebo Comparator): Placebo 1 tablet three times daily x 14 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Fasudil Hydrochloride — Fasudil 40 mg three times a day x 14 days
  Other Names: Fasudil
  Arms: Drug: Fasudil hydrochloride
Drug: Placebo Oral Tablet — Placebo oral tablet manufactured to mimic fasudil three times a day x 14 days
  Other Names: Placebo
  Arms: Drug: Placebo oral tablet

SUMMARY:
To evaluate the causal relationship between Rho/Rho kinase overactivity and mechanisms of vascular dysfunction in patients with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with >= 70% carotid stenosis (unilateral or bilateral) who are scheduled to undergo elective carotid endarterectomy
* Age >= 18 years
* Agreement of the operating surgeon for patient to participate

Exclusion Criteria:

* Surgery scheduled < 14 days after randomization
* Pregnancy
* ALT, GGT > 3x upper limit of normal (ULN)
* Creatinine > 3.5 mg/dL
* Prior intolerance to statins
* Reluctance to add or change dosage of statin therapy during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-03-13 (Actual); Primary Completion 2011-01-20 (Actual); Study Completion 2011-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anju Nohria, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: Fasudil: Fasudil 40 mg three times a day X 14 days
  Fasudil Hydrochloride: Fasudil 40 mg three times a day x 14 days
- Drug: Placebo: Placebo 1 tablet three times daily x 14 days
  Placebo Oral Tablet: Placebo manufactured to mimic fasudil three times a day x 14 days
Period: Overall Study
Arm/Group | Drug: Fasudil | Drug: Placebo
Started | 2 (Investigators blinded to study drug assignment due to early termination of study) | 0
Completed | 2 (Investigators blinded to study drug assignment due to early termination of study) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Fasudil | Drug: Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Rho/ROCK Expression With Concordant Increase in eNOS Expression/Activity in Carotid Specimens.
Description: We were going to compare Rho/ROCK expression and eNOS expression/activity in carotid specimens obtained from patients treated with fasudil and compare those to specimens obtained from patients treated with placebo. We anticipated that Rho/ROCK expression and activity would be decreased in spcimens obtained from fasudil treated patients compared to specimens obtained from patients treated with placebo. We also anticipated that eNOS expression and activity would be increased in specimens obtained from patients treated with fasudil compared to specimens obtained from patients treated with placebo.
Time Frame: >= 2 weeks
Arm/Group | Drug: Fasudil Hydrochloride | Drug: Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Drug: Fasudil | Drug: Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated early due to poor enrollment. The patients and physicians remained blinded to study drug assignment for the 2 patients who completed the protocol and no analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No